CLINICAL TRIAL: NCT03998813
Title: Chronic Pain and Functional Prognosis After Total Knee Replacement: Continuous Locoregional Analgesia by Catheter to the Femoral Triangle Versus Tissue Infiltration as Part of an Improved Rehabilitation After Surgery Approach
Acronym: TKAFTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHD038-19
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Knee Pain Chronic
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Locoregional analgesia by femoral triangle catheterization (Experimental)
  Interventions: Drug: Ropivacaine
- Tissue infiltration (Active Comparator)
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — Locoregional analgesia by femoral triangle catheterization
  Arms: Locoregional analgesia by femoral triangle catheterization
Drug: Ropivacaine — Tissue infiltration
  Arms: Tissue infiltration

SUMMARY:
The prevalence of Chronic Post-Surgical Pain (CPSP) after knee replacement, defined as pain greater than or equal to 4/10 on the visual analogue scale after the third postoperative month, is recognised as high, with an average of 20% (extremes of 7 to 45%).

These CPSP, when present, cause poor long-term joint functional prognosis and impaired quality of life for patients. Many predictive, pre-, per- and post-operative factors of these CPSP have been identified in recent years. The most common postoperative risk factor found in the literature is the intensity of early pain.

The treatment protocols for this early post-surgical pain are currently and mainly multimodal in nature, combining systemic analgesics (paracetamol, NSAIDs, morphine, gabapentins) and local anaesthetics, administered either in the form of peripheral nerve blocks (continuous or single injection) or in the form of tissue infiltration (TI) performed by the surgeon during the operation.

Very few of these techniques have been evaluated for their ability to reduce the incidence of CPSP. Drugs with antihyperalgesic properties such as ketamine or nefopam have been shown to be of no interest, except to reduce the proportion of pain of a neuropathic nature. Only the continuous femoral block has shown, to date, an interest in IT to reduce the incidence of these CPSP.

The main objective of this study is to show that a multimodal analgesia protocol based on continuous locoregional analgesia by femoral triangle catheterization could reduce the incidence of chronic post surgical pain compared to a protocol based on tissue infiltration.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient;
* Placement of unilateral tricompartmental knee prosthesis for gonarthrosis;
* ASA score between I and III ;
* Nonseptic scheduled surgery;
* Knee replacement scheduled on one of the first 3 days of the week (Monday to Wednesday included) in order to benefit from a homogeneous postoperative physical therapy;
* Able to understand the protocol;
* Having agreed to participate in the study and having given express oral consent;
* Affiliated with a social security system;
* Possibility of being followed as part of the protocol.

Exclusion Criteria:

* Age >= 86 years old;
* BMI > 35 ;
* Revision of knee replacement;
* Symptomatic contralateral osteoarthritis;
* Anterior of surgery on the operated knee (excluding arthroscopy and meniscectomy);
* Vascular surgery on the femoral vessels on the operated side;
* Concept of diffuse polyalgia syndrome (fibromyalgia);
* Documented neuropathy of the lower limb;
* Localized infection at the catheter puncture site (femoral triangle);
* Known allergy to Ropivacaine;
* Renal insufficiency (Clearance - CKD-EPI formula - creatinine <30 ml/min) and/or severe hepatic insufficiency (prothrombin blood level <50%) ;
* Inflammatory rheumatic disease (rheumatoid arthritis, ankylosing spondylitis...) ;
* Patients on immunosuppressive or systemically administered corticosteroid therapy;
* Daily use of level II or III analgesics for more than one month pre-operatively;
* Known intolerance to tier III analgesics;
* Allergy or contraindications to standard treatments administered per and postoperatively (paracetamol, NSAIDs);
* Patient undergoing knee surgery in the year prior to inclusion and participating in the study;
* Patients who do not cooperate or do not understand French, difficulties in understanding and evaluating the pain score, preoperative cognitive dysfunction making the interview unreliable;
* Patient under guardianship, curators, deprivation of liberty;
* Patient already engaged in another interventional clinical study (category 1);
* Pregnant or breastfeeding women, or women in a position to procreate who refuse an effective means of contraception;
* Refusal to participate;
* Inability to understand the protocol and its requirements, and/or to give express oral consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2024-04-08 (Actual)

PRIMARY OUTCOMES:
A walking pain assessment scale greater than or equal to 4 | Three months from the intervention
  Self-assessment scale to quantify the patient's pain on a virtual scale from 0 (no pain) to 10 (maximum pain imaginable)

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme GUILLEY, Study Director — CHD Vendée
Locations (5):
- France (5):
  - Clinique Victor PAUCHET, Amiens
  - Centre Hospitalier de Béthune Beuvry, Béthune
  - Centre Hospitalier Départemental Vendée, La Roche-sur-Yon
  - Hôpital des Diaconesses Croix Saint Simon, Paris
  - Hôpital Privé Sévigné, Rennes